CLINICAL TRIAL: NCT02164669
Title: Exploration of Neuroimaging and Biochemical Prognostic Indicators for Post-operative Cognitive Dysfunction After Coronary Artery Bypass Graft
Brief Title: Exploration of Neuroimaging and Biochemical Prognostic Indicators for POCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: wangqiang (Other)
Responsible Party: Sponsor-Investigator, wangqiang, Professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: 20130225-8
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Cognitive Dysfunction; Cognitive Impairment
Keywords: Inflammation; Coronary artery bypass graft; Magnetic Resonance Imaging
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognitive Dysfunction; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — 4ml venous blood will be collected, and serum IL-6， IL-8，TNF-α，NSE，S100β will be detected.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Postoperative cognitive dysfunction (POCD) may lead to serious consequences. But the underlying mechanisms are still unclear. Blood Oxygen Level Dependent (BOLD) fMRI and biochemical indicators will be used to explore the underlying mechanisms and represent a promising precursory target for diagnosis and treatment of POCD.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is one of the most common complications in patients undergoing cardiac surgery. POCD will not only increase the incidence of complications and mortality, but also influence the quality of life after discharging from the hospital. Many factors are associated with POCD, such as neuroinflammation, age, anesthetics, surgery stress response and genetic factors. But the underlying mechanisms are still unclear. Blood Oxygen Level Dependent (BOLD) fMRI, which could monitor the peripheral neuron spontaneous activity according to the ratio of oxyhemoglobin and deaeration hemoglobin in blood, will be used to investigate whether POCD is induced by the variance in neurons metabolism and spontaneous activity in brain regions. Meanwhile, biochemical indicators will be detected to explore the prompting indicators of POCD. The present study is aimed to represent a promising precursory target for diagnosis and treatment of POCD, and provide novel evidence and insights on the brain changes induced by POCD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years old
* Underwent selective CABG surgery

Exclusion Criteria:

* History of central nervous system or psychiatric disorders
* History of taking sedative, antidepressants, or alcoholism
* MMSE score less than 23
* Visual or auditory disorders
* Educated less than 7 years
* Claustrophobia
* Can not be supine
* Can not tolerate iodinated contrast agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will selective undergo Coronary Artery Bypass Grafting (CABG) surgery. Health adult
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The brain structure changes | 7 days postoperatively
  Using BOLD fMRI to investigate the variance of mean diffusivity and FA in nerve conduction bundle

SECONDARY OUTCOMES:
Mini-Mental State Examination | preoperative and 7 days, 3 months and 1 years postoperative
  Application of digital depth and breadth to test digital sign test Tracking the attachment test and assess depression self rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, MD, PhD, Study Director — Xijing Hospital; Zijun Gao, Dr., Principal Investigator — Xijing Hospital
Locations (1):
- Xijign Hospital, Xi'an, Shaanxi, China